CLINICAL TRIAL: NCT05603520
Title: Phenotyping Heterogeneity and Regionality of the Aorta
Acronym: PHaRAo
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: PHaRAo
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Large Artery Stiffness; Aortic Disease; Aortic Stenosis; Aortic Aneurysm
Keywords: aortic disease; large artery stiffness; aortic stenosis; aortic aneurysm
MeSH Terms: conditions — Aortic Diseases; Aortic Valve Stenosis; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — prospectively defined blood sampling protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers
  Interventions: Other: Collection of Clinical Data
- patients with aortic stenosis
  Interventions: Other: Collection of Clinical Data
- patients with aortic aneurysms
  Interventions: Other: Collection of Clinical Data

INTERVENTIONS:
Other: Collection of Clinical Data — prospectively and systematically collection of clinical research data from apparently healthy volunteers and patients with aortic stenosis and aneurysms

SUMMARY:
The aorta distributes cardiac stroke volume into the whole body through its finetuned conductance function, that is propagation and modulation of flow pattern. Physicomechanic properties of the aortic wall assure continuous and homogenous blood flow distribution to organs. The physicomechanic properties of the aortic wall are heterotopic: The collagen/elastin ratio doubles in the abdominal aorta as compared to the thoracic aorta. Malfunction of aortic conduction due to large artery stiffening (LAS) leads to premature wave reflection and excess pulsatility which translate into organ damage in low-resistance beds. The regional heterogeneity of aortic physicomechanic properties and their histomorphological substrate leading to altered regional hemodynamics are not well investigated.

Within the PHaRAo population, there is a spectrum of higher and lower risk patients. The aim of this cohort study is to collect prospectively and systematically clinical research data from PHaRAo patients. This cohort study is an open-end observational study to identify master switches in aortic disease

ELIGIBILITY:
1. apparently healthy volunteers

   Inclusion Criteria:

   • Healthy volunteers

   Exclusion Criteria:
   * < 18 years
   * Active Medication
   * Cardiovascular Disease
   * MRI not possible
2. Patients with Aortic Stenosis

   Inclusion Criteria:

   • Patients suffering from 3rd drgree Aortic Stenosis

   Exclusion Criteria:
   * < 18 years
   * MRI not possible
3. Patients with Aortic Aneurysms

Inclusion Criteria:

• Patients suffering from Aortic Aneurysms

Exclusion Criteria:

* < 18 years
* MRI not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers, patients with aortic stenosis, patients with aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progressive accelerated Large Artery Stiffening | 5 years
  measured by CMR
Development of Aortic Aneurysm | 5 years
  measured by CMR
Progressive accelerated Large Artery Stiffening | 5 years
  measured by tonometry

SECONDARY OUTCOMES:
Diastolic Dysfunction | 5 years
  measured by CMR
Diastolic Dysfunction | 5 years
  measured by echocardiography
Ejection Rate and Ejection Time | 5 years
  measured by CMR
Ejection Rate and Ejection Time | 5 years
  measured by echocardiography
Flow encoded regional MRI metrics | 5 years
  measured by CMR

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Christine Quast, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Christine Quast, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quast C, Bonner F, Polzin A, Veulemans V, Chennupati R, Gyamfi Poku I, Pfeiler S, Kramser N, Nankinova M, Staub N, Zweck E, Jokiel J, Keyser F, Hoffe J, Witkowski S, Becker K, Leuders P, Zako S, Erkens R, Jung C, Flogel U, Wang T, Neidlin M, Steinseifer U, Niepmann ST, Zimmer S, Gerdes N, Cortese-Krott MM, Feelisch M, Zeus T, Kelm M. Aortic Valve Stenosis Causes Accumulation of Extracellular Hemoglobin and Systemic Endothelial Dysfunction. Circulation. 2024 Sep 17;150(12):952-965. doi: 10.1161/CIRCULATIONAHA.123.064747. Epub 2024 Jun 5. PMID 38836358